CLINICAL TRIAL: NCT04416035
Title: A Phase 3, Multicenter, Randomized and Double-Blind Study to Assess the Similarity in Efficacy and Safety Between TRS003 and China-approved Bevacizumab in Subjects With Advanced Nonsquamous NSCLC
Brief Title: A Study to Compare the Similarity in Efficacy and Safety Between TRS003 and China-approved Bevacizumab® in NSCLC
Acronym: NSCLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Teruisi Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS00303001
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Advanced Non-squamous Non-small-cell Lung Cancer
MeSH Terms: interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRS003 (Experimental): TRS003 will be administered at 15 mg/kg by IV infusion on Day 1 of each cycle (every 3 weeks, Q3W). Paclitaxel will be administered at a dose of 200 mg/m^2 by IV infusion Q3W on Day 1 of each cycle，carboplatin will be administered at an AUC 6 mg/mL/ min by IV infusion Q3W on Day 1 of each cycle. Each cycle is 3 weeks. Treatments will continue until disease progression, death, intolerable toxicity, withdrawal of consent, investigator decision, or completion of 4-6 cycles of therapy. Maintenance therapy may be given at the discretion of the patient's primary oncologist.
  Interventions: Biological: TRS003; Drug: Carboplatin; Drug: Paclitaxel
- China-approved Bevacizumab (Active Comparator): China-approved bevacizumab will be administered at 15 mg/kg by IV infusion on Day 1 of each cycle (every 3 weeks, Q3W). Paclitaxel will be administered at a dose of 200 mg/m^2 by IV infusion Q3W on Day 1 of each cycle and carboplatin will be administered at an AUC 6 mg/mL/min (the maximum dose capped at 900 mg) by IV infusion Q3W on Day 1 of each cycle. Each cycle is 3 weeks. Treatments will continue until disease progression, death, intolerable toxicity, withdrawal of consent, investigator decision, or completion of 4-6 cycles of therapy. Maintenance therapy may be given at the discretion of the patient's primary oncologist.
  Interventions: Biological: China-approved Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Biological: TRS003 — TRS003 will be administered at 15 mg/kg by IV infusion on Day 1 of each cycle (every 3 weeks, Q3W). Each cycle is 3 weeks.
  Arms: TRS003
Biological: China-approved Bevacizumab — China-approved bevacizumab will be administered at 15 mg/kg by IV infusion on Day 1 of each cycle (every 3 weeks, Q3W).Each cycle is 3 weeks.
  Arms: China-approved Bevacizumab
Drug: Carboplatin — Carboplatin will be administered at an AUC 6 mg/mL/ min (the maximum dose capped at 900 mg) by IV infusion (over 15 - 30 minutes) Q3W on Day 1 of each cycle.
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 200 mg/m^2 by IV infusion (over 3 hours) Q3W on Day 1 of each cycle

SUMMARY:
This is a double-blind Phase 3 clinical trial evaluating the efficacy and safety of TRS003 and paclitaxel-carboplatin versus China-approved bevacizumab and paclitaxel-carboplatin in patients with unresectable, locally advanced, or metastatic non-squamous non-small cell lung cancer (NSCLC). Approximately 608 patients will be enrolled in this study from America, Europe, and Asia. Patients who sign the informed consent and meet the inclusion criteria, will be randomized (1:1) to receive either TRS003 in combination with paclitaxel and carboplatin or China-approved bevacizumab in combination with paclitaxel and carboplatin for 4 to 6 cycles.

DETAILED DESCRIPTION:
This is a randomized, double-blind, multinational, multicenter, active-control, parallel two-group Phase 3 clinical trial evaluating the efficacy and safety of TRS003 plus paclitaxel-carboplatin versus China-approved bevacizumab plus paclitaxel-carboplatin in patients with unresectable, locally advanced, recurrent or metastatic non-squamous NSCLC. Approximately 608 subjects will be enrolled into this study from America, Europe and Asia. Patients who sign the informed consent and meet the inclusion criteria will be randomized (1:1) to receive either TRS003 or China-approved bevacizumab in combination with paclitaxel-carboplatin for 4 to 6 cycles. Patients will be stratified by region (Asia, Europe and America), gender, and cigarette smoking habit (previous smoker, smoker and non-smoker).

Patients will receive either TRS003 (Arm A), or China-approved bevacizumab (Arm B) first followed by the administration of paclitaxel and carboplatin. TRS003 or China-approved bevacizumab will be administered at 15 mg/kg by intravenous (IV) infusion on Day 1 of each cycle (every 3 weeks, Q3W). Paclitaxel will be administered at a dose of 200 mg/m^2 by IV infusion (over 3 hours) Q3W on Day 1 of each cycle and carboplatin will be administered at an area under the plasma concentration-time curve (AUC) 6 mg/mL/ min (the maximum dose capped at 900 mg) by IV infusion (over 15 - 30 minutes) Q3W on Day 1 of each cycle. Each cycle is 3 weeks. Treatments will continue until disease progression, death, intolerable toxicity, withdrawal of consent, investigator decision, or completion of 4-6 cycles of therapy. Maintenance therapy may be given at the discretion of the patient's primary oncologist.

Efficacy will be evaluated by the investigator per RECIST v1.1 (Eisenhauer et al., 2009). Efficacy evaluation will be performed at baseline and every 6 weeks ± 7 days during the 4-6 cycle combination treatment periods. After completion of combination treatments, efficacy evaluations will be performed every 9 weeks ± 7 days (if patients received maintenance therapy). The analysis of Investigator-determined objective response rate (ORR) (RECIST v1.1) will be based on information obtained prior to Week 19. Investigator-determined duration of response (DOR) and progression-free survival (PFS) will also be evaluated according to RECIST v1.1. Data on overall survival (OS) will be collected. Central radiology review will not be required. However, for the purpose of quality control, the Sponsor may elect to have some or all tumor assessments to be reviewed by an independent imaging vendor.

Safety will be evaluated throughout the study. Adverse events will be recorded from the time of informed consent. Safety will be assessed based on periodically physical examination findings, vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, laboratory variables (hematology, coagulation tests, serum chemistries, urinalysis and pregnancy tests), and electrocardiogram (ECG) findings. Adverse events and laboratories will be graded according to National Cancer Institute (NCI) CTCAE v5.0.

Immunogenicity will be assessed in all patients who received at least one dose of TRS003 or China-approved bevacizumab. Samples will be assessed for the development of antidrug antibodies to either TRS003, or China-approved bevacizumab. Neutralizing antibodies (NAb) will assessed in samples that are antidrug antibody (ADA) positive. Trough pharmacokinetics (PK) samples will be collected and will be analyzed for interpretation of immunogenicity data and exploratory analysis when needed.

ELIGIBILITY:
Inclusion Criteria :

1. Male or female ≥ 18 years.
2. Signed and dated informed consent form.
3. Willing and able to comply with all study procedures.
4. Histologically or cytologically confirmed unresectable, locally advanced, recurrent, or metastatic nonsquamous NSCLC; if the tumor shows multiple histologies, the main cellular phenotype will be used. Must provide archived tumor tissue obtained within 3 years for epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) testing. If archival tissue meeting this requirement is not available, patients will undergo biopsy to be eligible for study entry.
5. No previous systemic therapy targeting the primary tumor or sites of metastases. Adjuvant therapy should be completed at least 6 months prior to study entry. Patients may have received radiation therapy if this was completed at least 1 month prior to entry and if other sites of measurable disease (per RECIST v11) are present.
6. At least one measurable lesion per RECIST v1.1.
7. ECOG performance status score 0 or 1.
8. Life expectancy ≥ 6months.
9. Adequate hepatic function as evidence by meeting all the following requirements:

   1. Total bilirubin ≤ 1.5 × upper limit of normal (ULN).
   2. Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 3×ULN or ALT ≤ 5 × ULN if liver metastases are present.
10. Adequate renal function as evidence by meeting all the following requirements:

    1. Serum creatinine ≤ 1.5 × ULN and calculated creatinine clearance (CrCL) > 50 mL/min (Cockroft-Gault Equation) or estimated glomerular filtration rate (GFR) > 50 mL/min.
    2. Urine dipstick for proteinuria < 2+. If urine dipstick is greater than or equal to 2+, proteinuria must be less than 2 g in 24 hours or the urine protein/creatinine ratio < 2.
11. Hematological function defined as:

    1. Platelet count ≥ 100,000/μl without transfusion within 2 weeks prior to the study screening.
    2. Prothrombin time, international normalized ratio or activated partial thromboplastin time < 1.5 × ULN.
    3. Absolute neutrophil count ≥ 1,500/μl without any medical interventional treatment within two weeks prior to the study screening (ie, granulocyte-colony stimulating factors and/or herbal remedies).
    4. Hemoglobin (Hb) ≥ 9 g/dl without the need for transfusion within 2 weeks prior to the study screening.

Exclusion Criteria ：

1. Known sensitizing EGFR mutations or ALK rearrangements.
2. Squamous lung cancer, mixed small cell and non-small cell lung cancer or squamous cell-dominant adeno-squamous lung cancer.
3. Tumor cavitation, invading into large blood vessels or close to large vessels (such as pulmonary artery or Superior vena cava.
4. Significant thrombotic or hemorrhagic events within 6 months prior to the study screening e.g., hemoptysis > 2.5 mL of red blood, gastrointestinal bleeding, hematemesis, central nervous system hemorrhage, severe epistaxis or vaginal bleeding, etc.
5. Severe cardiovascular disease, including cerebrovascular accident (CVA), transient ischemic attack (TIA), myocardial infarction and significant vascular disease (including but not limited to aneurysm requiring surgical repair or recent artery thrombosis); unstable angina pectoris, New York Heart Association (NYHA) class III or IV heart failure and uncontrollable arrhythmia within 6 months prior to entry.
6. History of active gastroduodenal ulcer, abdominal fistula as well as non-gastrointestinal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to the study screening.
7. Central nervous system (CNS) metastases; Subjects with asymptomatic CNS metastases who are neurologically stable ≥ 4 weeks following CNS-directed therapy with no evidence of CNS disease progression ≥ 4 weeks, and on a stable or decreasing dose of corticosteroids may be eligible and should be discussed with the Medical Monitor.
8. Concurrent malignancy within 5 years other than adequately treated primary cervical cancer, skin-squamous or basal cell carcinomas, prostatic cancer following radical resection that does not require therapy, prostate cancer treated with active surveillance, ductal carcinoma in situ of the breast, or < T1 urothelial carcinoma.
9. Uncontrolled hypertension (systolic blood pressure >150 mmHg and diastolic blood pressure >100 mmHg at the study screening), or a history of hypertension crisis or hypertensive encephalophy.
10. Active hepatitis B or hepatitis C virus. Patients with evidence of infection with hepatitis B who have an undetectable viral load are eligible for study entry. Patients with evidence of infection with hepatitis C should have completed curative therapy.
11. Known to be positive for human immunodeficiency virus (HIV) and with an AIDS defining opportunistic infection within 12 months of study entry or a CD4 T cell count < 359 cells/μL.
12. Full dose anticoagulants, including oral or parenteral; Low dose anti-coagulation (not intended to achieve a therapeutic INR) for port patency is permitted. No Factor Xa inhibitors. No aspirin or other nonsteroidal anti-inflammatory drugs that can inhibit platelet within ten days prior to screening. No history of hemorrhagic or thrombotic disorders (e.g., hemophilia, protein C deficiency).
13. Thoracic radiotherapy within 4 weeks prior to screening or palliative radiotherapy for metastasis outside thoracic region within 2 weeks prior to screening.
14. Any major surgical procedure within 28 days prior to screening or anticipated elective surgery during the study. Any minor surgery such as deep vein catheterization within 48 hours prior to the first dose of the study drugs.
15. Evidence of pericardial or pleural effusion or ascites that requires intervention.
16. Treatment history of monoclonal antibodies or small molecule inhibitors against vascular endothelial growth factor (VEGF) or its receptor (VEGFR), including bevacizumab.
17. Clinically uncontrolled active infection requiring systemic therapy within 2 weeks prior to entry.
18. Subject has known sensitivity to any of the products to be administered during the study, including mammalian cell derived drug products.
19. Participation in any other clinical trial within 4 weeks prior to screening. Recipient of any anticancer therapy (other than hormones used to treat breast cancer) within 4 weeks prior to screening.
20. Women of childbearing potential who are pregnant or is breast feeding or who do not consent to use highly effective methods of birth control during treatment and for an additional 120 days after the last administration of the protocol specified treatment.
21. Men with a partner of childbearing potential who does not consent to use highly effective methods of birth control during treatment and for an additional 120 days after the last administration of the protocol specified treatment.
22. Any condition that the Investigator or primary physician believes may not be appropriate for participating the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2020-08-17 (Actual); Primary Completion 2021-10-21 (Estimated); Study Completion 2021-11-10 (Estimated)

PRIMARY OUTCOMES:
ORR,Objective Response Rate | 19 weeks
  Investigator-determined confirmed ORR by Week 19 per RECIST v1.1 will be determined in the intention-to-treat (ITT) population in each arm.

SECONDARY OUTCOMES:
PFS, Progression-free survival | 19 weeks
  PFS is defined as the time from randomization to Investigator-determined progressive disease (PD) or death due to any cause in the absence of documented PD.
OS, Overall survival | 19 weeks
  OS is defined as the time from randomization to death due to any cause and will be analyzed by Kaplan-Meier method.
DOR, Duration of response | 19 weeks
  DOR is defined as the time from the date of the first documentation of Investigator-determined response in patients with confirmed objective tumor response (complete response or partial response) to the first documentation of Investigator determined disease progression (PD) or to death due to any cause in the absence of documented PD.
Number of Participants with Treatment-Related Adverse Events (AEs) | 23 weeks
  AEs will be assigned to preferred term using MedDRA and graded according to CTCAE v5.0.
Number of Participants with Immunogenicity | 23 weeks
  ADA will be assessed in all patients. NAb will be assessed in samples that are ADA positive
AUC0-inf, Area Under the Serum Concentration Versus Time Curve (Time 0 to Infinity) | 23 weeks
  PK will only be analyzed for interpretation of immunogenicity data and exploratory analysis when needed.
AUC0-t, Area Under the Serum Concentration Versus Time Curve (Time 0 to t) | 23 weeks
  PK will only be analyzed for interpretation of immunogenicity data and exploratory analysis when needed.
Cmax, Maximum Drug Concentration | 23 weeks
  PK will only be analyzed for interpretation of immunogenicity data and exploratory analysis when needed.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Chinese Academy of Medical Sciences
Locations (11):
- China (11):
  - Anhui Provincial Center Hospital, Hefei, Anhui
  - Chinese Academy of Medical Sciences, Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - The Second Affiliated Hospital of Xingtai Medical College, Xingtai, Hebei
  - Wuhan Fourth Hospital, Wuhan, Hubei
  - The Second Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - FAW General Hospital of Jilin Province, Changchun, Jilin
  - Jinan Central Hospital, Jinan, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Fifth People's Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Nanchong Central Hospital, Nanchong, Sichuan